CLINICAL TRIAL: NCT01754831
Title: Fluoride Administered and Retained After Topical Fluoride Varnish
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Peter Milgrom, Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 41117
Record Dates: First submitted 2012-10-10; First posted 2012-12-21 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2016-05

CONDITIONS: Healthy
Keywords: children; fluoride varnish

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluoride varnish (Other): Topical fluoride
  Interventions: Device: Fluoride varnish

INTERVENTIONS:
Device: Fluoride varnish — Topical application of fluoride varnish on present teeth
  Other Names: Premier Enamel Pro

SUMMARY:
The specific aim of the study is to determine the excess urinary fluoride and its time course after administration of an application of Premier Enamel Pro Varnish to the teeth of 12-15 month old infants. From these data the investigators can estimate the bioavailable (more precisely the equivalent) dose of sodium fluoride and the peak serum fluoride concentration that will allow an estimate of the margin of safety of the procedure.

DETAILED DESCRIPTION:
Fluoride varnish painted on the teeth is the standard method dentists use to prevent tooth decay (cavities) in preschool children in the United States. Fluoride varnish is not FDA approved specifically for prevention of cavities, but dentists may legally use it for this purpose. We want to study how much fluoride appears in the urine after the painting procedure to improve our knowledge of how the varnish works and its safety. The fluoride varnish is being used for research purposes for this study by permission of FDA (IND #110869).

Premier Dental Product Company's Enamel Pro Varnish will be used. Up to six children aged 12-15 months will be enrolled in this study. We measured urinary fluoride for 5 hours after application of fluoride varnish to teeth. Baseline levels were measured on a separate day.

ELIGIBILITY:
Inclusion Criteria:

* consent obtained from parent or legal guardian of participant
* children aged 12 - 15 months
* at least 1 erupted tooth
* in general good health

Exclusion Criteria:

* known allergy to any drug, latex, nuts, or resin components or components of toothpaste/dental prophylaxis product
* participant has stomatitis or other oral conditions that preclude applying fluoride varnish comfortably

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Urinalysis for fluoride levels | 2 days
  We want to study how much fluoride appears in the urine after the painting procedure to improve our knowledge of how the varnish works and its safety.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Principal Investigator — University of Washington
Locations (1):
- UW Center for Pediatric Dentistry, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milgrom P, Taves DM, Kim AS, Watson GE, Horst JA. Pharmacokinetics of fluoride in toddlers after application of 5% sodium fluoride dental varnish. Pediatrics. 2014 Sep;134(3):e870-4. doi: 10.1542/peds.2013-3501. Epub 2014 Aug 18. PMID 25136045